CLINICAL TRIAL: NCT01238120
Title: A Phase II Study of the Effects of Physical Activity and Low-Dose Ibuprofen on Cognitive Function in Cancer Patients Undergoing Chemotherapy
Brief Title: The Effects of Physical Activity and Low-Dose Ibuprofen on Cognitive Function in Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michelle Janelsins, PhD, MPH, Associate Professor, University of Rochester
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 31416; K07CA168886 (NIH)
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Results first posted 2021-03-17 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Cancer-related Cognitive Difficulties
Keywords: Cancer; Cognitive difficulties
MeSH Terms: conditions — Neoplasms | interventions — Ibuprofen; Anti-Inflammatory Agents, Non-Steroidal; Exercise; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo and Home-Based Exercise (Active Comparator): 200mg placebo (taken twice a day at least 8 hours apart) for a period of 6 weeks and a progressive walking and resistance band exercise program called Exercise for Cancer Patient (EXCAP) for a period of 6 weeks.
  Interventions: Behavioral: Home-Based Exercise; Drug: Placebo
- Ibuprofen 200mg BID, Home-Based Exercise (Active Comparator): 200mg ibuprofen (taken twice a day at least 8 hours apart) and a progressive walking and resistance band exercise program called Exercise for Cancer Patient (EXCAP) for a period of 6 weeks.
  Interventions: Drug: Ibuprofen; Behavioral: Home-Based Exercise
- Placebo (Placebo Comparator): 200mg placebo (taken twice a day at least 8 hours apart) for a period of 6 weeks.
  Interventions: Drug: Placebo
- Ibuprofen 200 mg BID (Active Comparator): 200mg ibuprofen (taken twice a day at least 8 hours apart) for a period of 6 weeks.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — 200 mg BID and 8 hours apart
  Other Names: nonsteroidal anti-inflammatory drug
  Arms: Ibuprofen 200 mg BID; Ibuprofen 200mg BID, Home-Based Exercise
Behavioral: Home-Based Exercise — A progressive walking and resistance band exercise program called Exercise for Cancer patient (EXCAP) for a 6 week period
  Other Names: Exercise for Cancer Patients
  Arms: Ibuprofen 200mg BID, Home-Based Exercise; Placebo and Home-Based Exercise
Drug: Placebo — 200mg BID and 8 hours apart
  Other Names: Sugar Pill
  Arms: Placebo; Placebo and Home-Based Exercise

SUMMARY:
This research seeks to determine if a combination of low-dose ibuprofen along with a structured home-based walking and progressive resistance exercise program, EXCAP, will be effective in reducing cognitive difficulties among cancer patients receiving chemotherapy.

DETAILED DESCRIPTION:
To conduct a feasibility pilot to assess preliminary efficacy of a 6 week course of ibuprofen (200 mg BID with does 8 hours apart) and a structured home based walking/progressive resistance program, EXCAP, alone or together, on cognitive function and levels of inflammatory molecules among cancer patients receiving chemotherapy (beginning at cycle 2). If these interventions prove to be useful and have potential benefit, they could have a substantial impact on treating cognitive difficulties experienced by cancer patients as well as improve quality of life. Moreover, if there is an effect of these interventions on cognitive functioning and inflammation, we will gain more knowledge of a possible mechanism of chemotherapy-related cognitive difficulties.

ELIGIBILITY:
Inclusion Criteria:

* Must report cognitive difficulties of 3 or higher on a 0-10 scale
* Must provide informed consent
* Be able to read English
* Have a primary diagnosis of cancer
* Be able to swallow medication
* Women of child-bearing potential must not be pregnant or become pregnant during the 6 week study
* Agree not to take NSAIDs during the 6 week intervention period
* Be scheduled to receive at least 2 additional cycles of oral or IV chemotherapy over the 42-day study period.
* Must have the approval of their treating physician to begin the exercise program and receive the ibuprofen
* Must be over 18 years of age

Exclusion Criteria:

* Currently taking a consistent dosage of a NSAID at least 3 days a week for the last 3 months that is over 400mg daily
* Have an allergy to ibuprofen
* Be identified as in active or maintenance stage of exercise behavior as assessed by the single-item exercise stages of change short form
* have physical limitations that contraindicate participation in sub-maximal physiological fitness testing or a low to moderate home-based walking and progressive resistance program
* have a history of peptic ulcer disease within the last 12 months
* Diagnosed with a neurodegenerative disease
* Had a myocardial infraction within the past 6 months
* Patients with a neutropenic episode during the first cycle of chemotherapy or at high risk for a neutropenic episode during future chemotherapy cycles at the treating physicians discretion
* Have confirmed metastatic disease to the central nervous system
* Have been hospitalized for a major psychiatric illness within the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-11; Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle C Janelsins, Ph.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No
Overall study results will be presented to participants, faculty and staff at the University of Rochester Medical Center. tudy results will be presented at professional meetings and published

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 110 subjects were consented.
  Of those 110 subjects, 97 were randomized, 13 excluded.
  Of the 13 excluded, 7 were by the subject's request, 5 had a medical problem which rendered them ineligible, and 1 was a screening failure.
  Of the 97 subjects randomized, 11 participants were excluded.
  Of the 11 excluded, 9 were by the subject's request and 2 were lost to follow up.
  86 participants received the intervention and completed baseline assessments (Overall Study Table Below).
Period: Overall Study
Arm/Group | Placebo and Home-Based Exercise | Placebo | Ibuprofen 200mg BID, Home-Based Exercise | Ibuprofen 200 mg BID
Started (Randomized) | 25 | 23 | 25 | 24
Received Intervention and Completed Baseline Assessments | 21 | 22 | 22 | 21
Completed | 17 | 22 | 21 | 18
Not Completed | 8 | 1 | 4 | 6
Not completed — Withdrawal by Subject | 4 | 1 | 2 | 5
Not completed — Lost to Follow-up | 2 | 0 | 1 | 1
Not completed — Withdrawn due to Medical Problem | 2 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo and Home-Based Exercise | Placebo | Ibuprofen 200mg BID, Home-Based Exercise | Ibuprofen 200 mg BID | Total
Number analyzed (Participants) | 25 | 23 | 25 | 24 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.19 (10.52) | 54.95 (12.51) | 54.86 (11.86) | 50.29 (8.92) | 53.60 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 22 | 21 | 87
  Male | 3 | 1 | 3 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 25 | 23 | 24 | 23 | 95
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 0 | 0 | 6
  White | 20 | 22 | 24 | 23 | 89
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Cancer Type [Count of Participants; unit: Participants]
  Breast | 19 | 19 | 17 | 18 | 73
  Gastrointestinal | 4 | 4 | 7 | 5 | 20
  Other | 2 | 0 | 1 | 1 | 4
Education Level [Count of Participants; unit: Participants]
  Highschool/GED or less | 4 | 4 | 1 | 2 | 11
  2 to 4 Year Degree | 13 | 10 | 11 | 15 | 49
  Graduate Degree | 3 | 8 | 9 | 4 | 24
  Unknown | 5 | 1 | 4 | 3 | 13
Cancer Stage [Count of Participants; unit: Participants] — Stage 1.This stage is usually a small cancer or tumor that has not grown deeply into nearby tissues. It also has not spread to the lymph nodes or other parts of the body.
  Stage 2 and 3.These stages indicate larger cancers or tumors that have grown more deeply into nearby tissue. They may have also spread to lymph nodes but not other parts of the body.
  Stage 4.This stage means that the cancer has spread to other organs or parts of the body. It may also be called metastatic cancer.
  Stage 1 is best, Stage 4 is worst.
  Participants
    Stage 1 | 2 | 4 | 5 | 2 | 13
    Stage 2 | 11 | 7 | 6 | 9 | 33
    Stage 3 | 4 | 6 | 11 | 5 | 26
    Stage 4 | 8 | 6 | 3 | 8 | 25

OUTCOME MEASURES:

1. Primary Outcome: Memory Performance as Assessed by Computerized Cognitive Assessment - Mean Values by Arm
Description: Memory performances (percent correct across delays) as assessed by the objective CANTAB delayed matching to sample task Percentage correct range (0 to 100) Higher percentage is better
Time Frame: Baseline and 6 weeks
Population: Note: Whenever the 6-week number of subject is less than the baseline number of subject this is due to the data not being available. n=17 for Placebo and Home-Based Exercise (1-withdrawal by subject, 1-lost to followup, 2-withdrawal due to medical reason); n=22 for Placebo Only; n=21 for Ibuprofen and Home-Based Exercise (1-withdrawal due to medical reason ); n=18 for Ibuprofen Only (2-withdrawal due to subject, 1=lost to followup)
Measure: Mean (Standard Deviation); unit: % correct
Arm/Group | Placebo and Home-Based Exercise | Placebo | Ibuprofen 200mg BID, Home-Based Exercise | Ibuprofen 200 mg BID
Number analyzed (Participants) | 21 | 22 | 22 | 21
% correct
  Basline | 75.2 (19.9) | 82.7 (17.8) | 83.6 (19.2) | 74.3 (20.1)
  6 Weeks: number analyzed (Participants) | 17 | 22 | 21 | 18
  6 Weeks | 89.4 (10.3) | 90.0 (10.2) | 87.6 (16.1) | 90.0 (15.7)
Statistical Analysis 1: Comparison: Placebo and Home-Based Exercise vs Placebo vs Ibuprofen 200mg BID, Home-Based Exercise vs Ibuprofen 200 mg BID; Test type: Superiority; p = 0.9168, ANCOVA

2. Secondary Outcome: Cognitive Functioning Score as Assessed by FACT-COG Questionnaire - Perceived Cognitive Impairment (PCI) - Mean Values by Arm
Description: Cognitive functioning score as assessed subjectively by a psychometrically validated instrument (FACT-COG) - Perceived Cognitive Impairment (PCI) (min=0, max=116) Higher Score is better
Time Frame: Baseline and 6 weeks
Population: Note: Whenever the 6-week number of subjects or baseline number of subjects is less than the number reported per arm this is due to the data not being available. n=17 for Placebo and Home-Based Exercise (1-withdrawal by subject, 1-lost to followup, 2-withdrawal due to medical reason); n=22 for Placebo Only; n=20 for Ibuprofen and Home-Based Exercise (1-withdrawal due to medical reason, 1-unknown ); n=18 for Ibuprofen Only (2-withdrawal due to subject, 1=lost to followup)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo and Home-Based Exercise | Placebo | Ibuprofen 200mg BID, Home-Based Exercise | Ibuprofen 200 mg BID
Number analyzed (Participants) | 21 | 22 | 22 | 21
score on a scale
  Baseline: number analyzed (Participants) | 20 | 22 | 21 | 21
  Baseline | 74.7 (22.0) | 72.7 (18.1) | 85.9 (17.1) | 76.2 (18.9)
  6 Weeks: number analyzed (Participants) | 17 | 22 | 20 | 18
  6 Weeks | 80.5 (19.7) | 76.5 (20.2) | 88.0 (21.0) | 78.9 (21.8)
Statistical Analysis 1: Comparison: Placebo and Home-Based Exercise vs Placebo vs Ibuprofen 200mg BID, Home-Based Exercise vs Ibuprofen 200 mg BID; Test type: Superiority; p = 0.6536, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study intervention period. Approximately 6 weeks
Description: Adverse event definition does not differ from clinicaltrials.gov definition. A serious adverse event (SAE) is any adverse event, occurring at any dose and regardless of causality that: Results in death, Is life-threatening, Requires inpatient hospitalization or prolongation of existing hospitalization, Results in persistent or significant disability/incapacity, Is a congenital anomaly/birth defect, or is an important medical event.
Arm/Group | Placebo and Home-Based Exercise | Placebo | Ibuprofen 200mg BID, Home-Based Exercise | Ibuprofen 200 mg BID
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23 | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 3/25 | 0/23 | 0/25 | 1/24
Other Adverse Events (participants affected / at risk) | 2/25 | 6/23 | 10/25 | 3/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo and Home-Based Exercise (N=25) | Placebo (N=23) | Ibuprofen 200mg BID, Home-Based Exercise (N=25) | Ibuprofen 200 mg BID (N=24)
Infection - Urinary Tract (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Melena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis Media (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo and Home-Based Exercise (N=25) | Placebo (N=23) | Ibuprofen 200mg BID, Home-Based Exercise (N=25) | Ibuprofen 200 mg BID (N=24)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Puritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial Thrombus (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasm benign - Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sore Throat (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain - Postoperative (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/20/NCT01238120/Prot_SAP_000.pdf